CLINICAL TRIAL: NCT03698266
Title: Is Needle Knife Fistulotomy An Effective First Step Strategy For All ERCPs?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lawrence Charles Hookey (Other)
Responsible Party: Sponsor-Investigator, Lawrence Charles Hookey, Associate Professor, Medical Director - Endoscopy Unit, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DMED-2175-18
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: ERCP; Biliary Disease Tract; Biliary Disease
Keywords: Needle Knife Fistulotomy; Sphincterotomy; Post-ERCP pancreatitis
MeSH Terms: conditions — Biliary Tract Diseases; Gallbladder Diseases

STUDY DESIGN:
Intervention Model Description: All patients enrolled in the study will consent to a needle knife fistulotomy as a starting technique to gain access to the biliary system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Enrolled Patients (Other): Receive needle knife fistulotomy as a starting technique to gain access to the biliary system
  Interventions: Procedure: Needle knife fistulotomy

INTERVENTIONS:
Procedure: Needle knife fistulotomy — A needle knife fistulotomy uses a tiny knife to cut directly into the ampulla to gain access to the biliary system in patients undergoing ERCP

SUMMARY:
Participants in this study will be undergoing a procedure called an endoscopic retrograde cholangiopancreatography (ERCP). This procedure is most commonly performed to help treat conditions affecting specific areas of the digestive system called the pancreas and bile ducts.

Patients will consent to allow the study physician to access these areas of the digestive system by making a cut using a technique called a needle-knife fistulotomy. If the physician is unable to gain access through this method, they will make the cut using a technique called a sphincterotomy.

DETAILED DESCRIPTION:
The ERCP procedure enables doctors to examine the regions of the digestive system called the pancreas and bile ducts. After sedating a patient, a bendable tube with a light (called an endoscope), is inserted through the mouth and into the digestive system. Within the digestive system, the doctor is able to identify the opening to where the gallbladder drains into the small bowel called the ampulla. Using the endoscope, a small plastic tube is then placed in the opening and dye (also called contrast material) is injected bile duct (where bile leaves the liver from). X-ray pictures can then be taken to provide further information to the doctor.

Sometimes it is necessary to make a cut to enlarge the opening to allow easier removal of stones from the bile duct or to place plastic tubes (stents) in the bile duct. To make this cut, there are two different approaches that the doctor can take:

1. The standard way of making the cut is referred to as a "sphincterotomy". Using this method, a heated metal wire cuts the opening to the bile duct after a wire has been passed into it.
2. The second way of making the cut is referred to as a "pre-cut". There are various types of "pre-cut" techniques; the technique being evaluated in this study is called the "needle knife fistulotomy". When using this technique, the doctor makes a cut directly into the bile duct using a tiny knife called a "needle knife".

Currently, there is not a standard that tells doctors what cutting technique to use. The decision is entirely up to the individual doctor.

Patients that participate in this study give their permission to allow the study doctor to use the "needle knife fistulotomy" cutting technique first to gain access to the bile ducts. If the study doctor is unable to gain access through this method, then they will use the standard sphincterotomy technique.

The purpose of this study, called a feasibility study, is to determine if the needle-knife fistulotomy is at least as safe and effective as the standard access technique, if not safer.

If it can be shown that the needle-knife fistulotomy is safer and/or more effective, then it could change the way that doctors conduct this procedure in Canada and the rest of the world.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, ages > 18, with an intact sphincter undergoing ERCP by at Kingston Health Sciences Center for therapeutic purposes who can provide informed consent. This includes patients who have confirmed choledocholithiasis on imaging and those who have a high suspicion of it based on imaging and lab values. Patients with and without a high suspicion for cholangitis will be eligible for the study. Other indications include: type 1 sphincter of Oddi dysfunction, gallstone pancreatitis or other benign pancreaticobiliary duct diseases including strictures, primary sclerosing cholangitis and Mirizzi's syndrome. Furthermore, patients with suspected diagnosis of biliary leak following cholecystectomy will also be considered for enrollment in this study.
2. Ability to read and understand the English language

Exclusion criteria:

1. Bleeding disorder (Von Willebrand disorder, platelet count <100 000, or INR >1.5)
2. Therapeutic level anticoagulation with low molecular weight heparin (LMWH), warfarin, or a direct-acting oral anticoagulant (DOAC)
3. Prior biliary sphincterotomy
4. Altered upper GI tract anatomy (e.g. prior gastric bypass surgery such as Roux-en-Y or Billroth 2 gastrojejunostomy)
5. Evidence of Malignant infiltration of the ampulla or peri-ampullary area.
6. Inability to identify intra-duodenal portion of the bile duct, including deep peri-ampullary diverticulum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Post-ERCP pancreatitis | Up to 7 days post-procedure
  The primary objective to be examined is the incidence of post-ERCP pancreatitis

SECONDARY OUTCOMES:
Technical success | Day of procedure
  Determined by successful cannulation of the CBD as evidenced on cholangiogram

OTHER OUTCOMES:
Total procedure time | Day of procedure
  Measured for completed procedures from the time of esophageal intubation to the time of scope withdrawal from the patient mouth
Time to successful cannulation | Day of procedure
  Measured from the time of identification of the papilla to successful CBD cannulation as evident by the cholangiogram

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C Hookey, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robison LS, Varadarajulu S, Wilcox CM. Safety and success of precut biliary sphincterotomy: Is it linked to experience or expertise? World J Gastroenterol. 2007 Apr 21;13(15):2183-6. doi: 10.3748/wjg.v13.i15.2183. PMID 17465498
- [Background] Maydeo A, Borkar D. Techniques of selective cannulation and sphincterotomy. Endoscopy. 2003 Aug;35(8):S19-23. doi: 10.1055/s-2003-41532. PMID 12929049
- [Background] Kahaleh M, Tokar J, Mullick T, Bickston SJ, Yeaton P. Prospective evaluation of pancreatic sphincterotomy as a precut technique for biliary cannulation. Clin Gastroenterol Hepatol. 2004 Nov;2(11):971-7. doi: 10.1016/s1542-3565(04)00484-7. PMID 15551249
- [Background] Sherman S, Ruffolo TA, Hawes RH, Lehman GA. Complications of endoscopic sphincterotomy. A prospective series with emphasis on the increased risk associated with sphincter of Oddi dysfunction and nondilated bile ducts. Gastroenterology. 1991 Oct;101(4):1068-75. PMID 1889699
- [Background] Shakoor T, Geenen JE. Pre-cut papillotomy. Gastrointest Endosc. 1992 Sep-Oct;38(5):623-7. doi: 10.1016/s0016-5107(92)70537-9. No abstract available. PMID 1397929
- [Background] Foutch PG. A prospective assessment of results for needle-knife papillotomy and standard endoscopic sphincterotomy. Gastrointest Endosc. 1995 Jan;41(1):25-32. doi: 10.1016/s0016-5107(95)70272-5. PMID 7698621
- [Background] Huibregtse K, Katon RM, Tytgat GN. Precut papillotomy via fine-needle knife papillotome: a safe and effective technique. Gastrointest Endosc. 1986 Dec;32(6):403-5. doi: 10.1016/s0016-5107(86)71921-4. No abstract available. PMID 3803839
- [Background] Lopes L, Dinis-Ribeiro M, Rolanda C. Early precut fistulotomy for biliary access: time to change the paradigm of "the later, the better"? Gastrointest Endosc. 2014 Oct;80(4):634-641. doi: 10.1016/j.gie.2014.03.014. Epub 2014 May 6. PMID 24814775
- [Background] Testoni PA, Mariani A, Aabakken L, Arvanitakis M, Bories E, Costamagna G, Deviere J, Dinis-Ribeiro M, Dumonceau JM, Giovannini M, Gyokeres T, Hafner M, Halttunen J, Hassan C, Lopes L, Papanikolaou IS, Tham TC, Tringali A, van Hooft J, Williams EJ. Papillary cannulation and sphincterotomy techniques at ERCP: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2016 Jul;48(7):657-83. doi: 10.1055/s-0042-108641. Epub 2016 Jun 14. PMID 27299638
- [Background] ASGE Standards of Practice Committee; Chandrasekhara V, Khashab MA, Muthusamy VR, Acosta RD, Agrawal D, Bruining DH, Eloubeidi MA, Fanelli RD, Faulx AL, Gurudu SR, Kothari S, Lightdale JR, Qumseya BJ, Shaukat A, Wang A, Wani SB, Yang J, DeWitt JM. Adverse events associated with ERCP. Gastrointest Endosc. 2017 Jan;85(1):32-47. doi: 10.1016/j.gie.2016.06.051. Epub 2016 Aug 18. No abstract available. PMID 27546389
- [Background] ASGE Standards of Practice Committee; Chathadi KV, Chandrasekhara V, Acosta RD, Decker GA, Early DS, Eloubeidi MA, Evans JA, Faulx AL, Fanelli RD, Fisher DA, Foley K, Fonkalsrud L, Hwang JH, Jue TL, Khashab MA, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Sharaf R, Shaukat A, Shergill AK, Wang A, Cash BD, DeWitt JM. The role of ERCP in benign diseases of the biliary tract. Gastrointest Endosc. 2015 Apr;81(4):795-803. doi: 10.1016/j.gie.2014.11.019. Epub 2015 Feb 7. No abstract available. PMID 25665931
- [Background] Freeman ML, Guda NM. ERCP cannulation: a review of reported techniques. Gastrointest Endosc. 2005 Jan;61(1):112-25. doi: 10.1016/s0016-5107(04)02463-0. No abstract available. PMID 15672074
- [Background] Katsinelos P, Gkagkalis S, Chatzimavroudis G, Beltsis A, Terzoudis S, Zavos C, Gatopoulou A, Lazaraki G, Vasiliadis T, Kountouras J. Comparison of three types of precut technique to achieve common bile duct cannulation: a retrospective analysis of 274 cases. Dig Dis Sci. 2012 Dec;57(12):3286-92. doi: 10.1007/s10620-012-2271-8. Epub 2012 Jun 20. PMID 22714730
- [Background] Sundaralingam P, Masson P, Bourke MJ. Early Precut Sphincterotomy Does Not Increase Risk During Endoscopic Retrograde Cholangiopancreatography in Patients With Difficult Biliary Access: A Meta-analysis of Randomized Controlled Trials. Clin Gastroenterol Hepatol. 2015 Oct;13(10):1722-1729.e2. doi: 10.1016/j.cgh.2015.06.035. Epub 2015 Jul 2. PMID 26144018
- [Background] Cha SW, Leung WD, Lehman GA, Watkins JL, McHenry L, Fogel EL, Sherman S. Does leaving a main pancreatic duct stent in place reduce the incidence of precut biliary sphincterotomy-associated pancreatitis? A randomized, prospective study. Gastrointest Endosc. 2013 Feb;77(2):209-16. doi: 10.1016/j.gie.2012.08.022. Epub 2012 Oct 22. PMID 23084272
- [Background] Mariani A, Di Leo M, Giardullo N, Giussani A, Marini M, Buffoli F, Cipolletta L, Radaelli F, Ravelli P, Lombardi G, D'Onofrio V, Macchiarelli R, Iiritano E, Le Grazie M, Pantaleo G, Testoni PA. Early precut sphincterotomy for difficult biliary access to reduce post-ERCP pancreatitis: a randomized trial. Endoscopy. 2016 Jun;48(6):530-5. doi: 10.1055/s-0042-102250. Epub 2016 Mar 18. PMID 26990509
- [Background] Freeman ML. Precut (access) sphincterotomy. Techniques in Gastrointestinal Endosocpy. 1999;1(1):40-8.
- [Background] Ayoubi M, Sansoe G, Leone N, Castellino F. Comparison between needle-knife fistulotomy and standard cannulation in ERCP. World J Gastrointest Endosc. 2012 Sep 16;4(9):398-404. doi: 10.4253/wjge.v4.i9.398. PMID 23125897
- [Background] Jin YJ, Jeong S, Lee DH. Utility of needle-knife fistulotomy as an initial method of biliary cannulation to prevent post-ERCP pancreatitis in a highly selected at-risk group: a single-arm prospective feasibility study. Gastrointest Endosc. 2016 Nov;84(5):808-813. doi: 10.1016/j.gie.2016.04.011. Epub 2016 Apr 19. PMID 27102829
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Dumonceau JM, Andriulli A, Elmunzer BJ, Mariani A, Meister T, Deviere J, Marek T, Baron TH, Hassan C, Testoni PA, Kapral C; European Society of Gastrointestinal Endoscopy. Prophylaxis of post-ERCP pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - updated June 2014. Endoscopy. 2014 Sep;46(9):799-815. doi: 10.1055/s-0034-1377875. Epub 2014 Aug 22. PMID 25148137
- [Result] Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996 Sep 26;335(13):909-18. doi: 10.1056/NEJM199609263351301. PMID 8782497